CLINICAL TRIAL: NCT04407299
Title: Impact of COVID-19 Pandemic on Attitude, Behaviour and Mental Health of Patients With Rheumatic Diseases
Brief Title: COVID-19 Impact on Rheumatic Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mervat Eissa, Associate Prpfessor, Cairo University
Other Study IDs: COVID-19Rheum
Record Dates: First submitted 2020-05-23; First posted 2020-05-29 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: COVID
Keywords: Rheumatic patients; COVID-19; behaviour; Mental health
MeSH Terms: conditions — COVID-19; Behavior; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: 180 patients diagnosed with autoimmune rheumatic disease. Patients are RA SLE Rhupus AS Behcet Sjogren Vasculitis FM Polymyalgia APA Sarcoidosis IBD Scleroderma DM PSA Mixed
  Interventions: Behavioral: self-administered structured questionnaire
- 2: control group composed of 180 healthy individuals (matched for age and sex)
  Interventions: Behavioral: self-administered structured questionnaire

INTERVENTIONS:
Behavioral: self-administered structured questionnaire — It was designed as a self-administered questionnaire with closed questions (yes/no questions, rating scale and multiple choice questions) and some open ended questions.

SUMMARY:
A study to assess the impact of coronavirus disease 2019 (COVID-19) pandemic on the attitude, behaviour and mental health of rheumatic patients and to compare them with healthy individuals.

DETAILED DESCRIPTION:
To assess the impact of coronavirus disease 2019 (COVID19) pandemic on the attitude, behaviour and mental health of rheumatic patients and to compare them with healthy individual. This is cross-sectional survey, 360 participants were included and divided into cases group composed of 180 patients with rheumatic diseases and control group composed of 180 healthy people. Data were collected via a self-administered structured questionnaire (Google form) which was sent to participants via social networks and emails to different rheumatic patients and healthy individuals. Mental health was measured by the five-item Brief Symptom Rating Scale (BSRS-5).

Conclusion: Mental health should be addressed in the same manner we deal with the infectious disease itself, being of no less importance. It is essential for mental health professionals provide psychological support to vulnerable populations, including the infected and chronically ill patients and their families, individuals, communities and health care workers.

ELIGIBILITY:
Inclusion Criteria:

* adult patient with diagnosed rheumatic disease

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: a total of 360 participants were included in this study and divided into two groups: cases group composed of 180 patients with rheumatic diseases and control group composed of 180 healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Score of five-item Brief Symptom Rating Scale (BSRS-5) | 3 weeks
  7. Six questions for mental health assessment for patients and controls: Mental health was measured by the five-item Brief Symptom Rating Scale (BSRS-5) which was derived from the 50-item BSRS

CONTACTS AND LOCATIONS:
Overall Officials: Mervat Eissa, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy Hospital, Cairo, Non-US/Non-Canadian, Egypt

IPD SHARING:
Plan to Share IPD: No